CLINICAL TRIAL: NCT06341959
Title: Can a Low-threshold Check-up Motivate Older People to Schedule a Dental Visit? A Randomized Controlled Trial
Brief Title: Can a Low-threshold Check-up Motivate Older People to Schedule a Dental Visit?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GerodentPLUS1
Record Dates: First submitted 2024-02-06; First posted 2024-04-02 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Oral Disease
MeSH Terms: conditions — Mouth Diseases | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: The intervention group will be provided with tools to facilitate dental contact and will be informed about the importance of regular dental visits. Participants are given the opportunity to receive an oral examination. Afterwards, each participant will receive brochures with oral hygiene instructions to take home. Participants will receive information about any identified oral pathology. A referral letter for the dentist and a report for the general practitioner will also be prepared to increase social influence. If the participant doesn't have a dentist, the participant will receive a list of contact information for dentists in the area.
  In the control group, no oral examination will be performed. However, participants will be given a list of nearby dentists and flyers with oral hygiene instructions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will be provided with tools to facilitate dental contact and will be informed about the importance of regular dental visits. Participants are given the opportunity to receive an oral examination. Afterwards, each participant will receive brochures with oral hygiene instructions to take home. Participants will receive information about any identified oral pathology. A referral letter for the dentist and a report for the general practitioner will also be prepared to increase social influence. If the participant doesn't have a dentist, the participant will receive a list of contact information for dentists in the area.
  Interventions: Procedure: Oral screening
- Control Group (No Intervention): In the control group, no oral examination will be performed. However, participants will be given a list of nearby dentists and flyers with oral hygiene instructions.

INTERVENTIONS:
Procedure: Oral screening — The participants in the intervention group will receive an oral examination. Subsequently, information about any identified problem will be given. Lastly, participants will receive a referral letter for their dentist and a report for the general practitioner. If the participants don't have a regular dentist, they will also be given a list with contact information of dentists in the area.
  Arms: Intervention Group

SUMMARY:
There is little research on the effect of oral screening campaigns for improving oral health in older people. Therefore, the aim of this study is to investigate the effect of a low-threshold contact with an oral health professional, including an oral health examination, on dental attendance of older people (65 years of age or older).

DETAILED DESCRIPTION:
The intervention group will be provided with tools to facilitate dental contact and will be informed about the importance of regular dental visits. Participants are given the opportunity to receive an oral examination. Afterwards, each participant will receive brochures with oral hygiene instructions to take home. Participants will receive information about any identified oral pathology. A referral letter for the dentist and a report for the general practitioner will also be prepared to increase social influence. If the participant doesn't have a dentist, the participant will receive a list of contact information for dentists in the area.

In the control group, no oral examination will be performed. However, participants will be given a list of nearby dentists and flyers with oral hygiene instructions.

In this way, we want to find out whether the presence of a dental professional with tailored advice is crucial to motivate an elderly person to good oral care.

ELIGIBILITY:
Inclusion criteria:

* 65 years of age or older
* home-dwelling within the selected regions (ELZ RITS en ELZ Scheldekracht)
* Dutch speaking
* no dental check-up in the last 12 months
* sufficient cognitive ability to answer the questions

Exclusion criteria:

- Failure to meet inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Contacted a dentist | 4 months
  Number of participants that have contacted a dentist within 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Janssens, Principal Investigator — University Ghent
Locations (1):
- UGent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
Privacy of the participants

REFERENCES:
- [Derived] De Vleeschauwer A, Poppe L, Colman R, Janssens B. Can a low-threshold check-up motivate older adults to schedule a dental visit? Study protocol for a randomized controlled trial. Trials. 2025 Jan 20;26(1):23. doi: 10.1186/s13063-025-08728-7. PMID 39833951

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT06341959/Prot_SAP_ICF_000.pdf